CLINICAL TRIAL: NCT03719274
Title: Minimally Invasive Non-surgical Vitamin C Injection Versus the Conventional Surgical Depigmentation in Treatment of Gingival Hyperpigmentation of the Anterior Esthetic Zone: Prospective Study
Brief Title: Vitamin C Depigmenattion Versus Conventional Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, nermin mohammed ahmed yussif, assistant lecturer, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Melanin Hyperpigmentation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non-surgical vitamin c depigmentation (Experimental): locally injected vitamin c is used to depigment the hyperpigmented gingival tissues
  Interventions: Dietary Supplement: vitamin c depigementation
- surgical depigmentation (Active Comparator): the conventional scalpel surgical technique is used to depigment the hyperpigmented gingival tissues
  Interventions: Dietary Supplement: vitamin c depigementation

INTERVENTIONS:
Dietary Supplement: vitamin c depigementation — locally injected vitamin c depigementation

SUMMARY:
Although physiologic gingival hyperpigmentation is not a pathologic condition, it is considered one of the main esthetic problems in dentistry. It was found that the attached gingiva is the most frequently pigmented intraoral tissues followed by the papillary gingiva and the alveolar mucosa

DETAILED DESCRIPTION:
In addition to all of the previously mentioned actions of vitamin C, it was found to be involved in depigmentation due to several factors that not only depend on its direct effect on melanin and melanocytes but also due to the overall effect on the applied tissues. Melanin is one of the main reservoir for ROS, copper and calcium in the tissue cells . Once vitamin C is introduced to the target tissue, it binds efficiently to melanin due to the ROS, calcium and copper content which causes intracellular deficiency of these items and the inability of the cells to produce melanin. Calcium deficiency causes failure of melanocytes to perform cellular adhesion to keratinocytes as calcium is essential to form cadherins . Adhesion to keratinocytes is important stimulator to melanocytes in order to produce melanin, format dendrites and transfer the produced melanin to neighboring cells . Shortage of the intercellular copper limits the formation of tyrosin, tyrosinase enzyme and peroxidase enzyme which in turn stops the melanin production .

Therefore, the aim of the present study is to compare the clinical efficiency of the non-surgical intraepidermal injection of vitamin C in comparison to the gold standard surgical technique (scalpel technique) for gingival depigmentation.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-50 y
* medically free;
* physiologic gingival hyperpigmentation related to esthetic region were selected.

Exclusion Criteria:

All the reasons that could provoke an inflammatory reaction were excluded such as:

* systemic diseases (especially auto-immune diseases and chemotherapy uptake);
* pregnant and lactating mothers;
* usage of chlorhexidine or povidone iodine;
* Local causes (smoking and periodontitis).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
gingival color change | 6 months
  the degree of gingival color is determined by 2 different color indices

CONTACTS AND LOCATIONS:
Overall Officials: nermin yussif, Study Director — msa university

IPD SHARING:
Plan to Share IPD: Undecided